CLINICAL TRIAL: NCT04905966
Title: Effect of a Physical Activity and Nutrition Education Intervention on Obesity Prevalence in Schoolchildren From Caaguazu Department, Paraguay: A Clustered Randomized Controlled Trial
Brief Title: Effect of a Physical Activity and Nutrition Education Intervention on Obesity Prevalence in Schoolchildren
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patricia Celestina Ríos Mujica (Other)
Collaborators: PROCIENCIA, Consejo Nacional de Ciencia y Tecnología (Unknown)
Responsible Party: Sponsor-Investigator, Patricia Celestina Ríos Mujica, Field Coordinator, Instituto Regional de Investigación en Salud "Kaneo Shibata" UNCA
Organization: Instituto Regional de Investigación en Salud "Kaneo Shibata" UNCA (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PINV15426
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Childhood Obesity
Keywords: Childhood Obesity, Nutrition Education, Physical Activity; Intervention, Schools
MeSH Terms: conditions — Pediatric Obesity; Motor Activity | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Four groups of participants received four different interventions: (1) Nutrition education + Physical Activity; (2) Control
Who Masked: Participant
Masking Description: Three lists of schools were built, according to type of institution and area where the school is located. The first list corresponded to rural public schools, the second to urban public schools and the last to urban private schools.
  Each of the lists contained the type of institution (public / private), the area where it is located (urban / rural), the name of the school and the district to which it belongs. The schools were masked with an identifier number in order to avoid bias during the assignment to the groups (intervened / control). Schools were selected using a computer based list (...)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition education + Physical activity intervention (Experimental): Physical Activity and Nutrition Education: An additional 45 minute weekly physical education class and 5 weekly active break sessions of 10 minutes each will be added to the provisions of the children's curriculum. In addition, schools will receive high intensity nutrition education, that is, 3 weekly nutrition education classes of one hour in each session over a period of 6 months.
  Interventions: Behavioral: Nutrition education and Physical activity intervention
- Control (No Intervention): Schools receiving a lower intensity nutrition education served as control. This group received 3 sessions of 1 hour with a total of 3 educational sessions over the 6 month period. The educational material was the same as the intervention group but the development of lessons was not as specific and deep as the intervention group.

INTERVENTIONS:
Behavioral: Nutrition education and Physical activity intervention — Schools randomized to the experimental group received nutrition education sessions and physical activity classes.
  Arms: Nutrition education + Physical activity intervention

SUMMARY:
Childhood obesity is a major global public health problem. Several strategies have been implemented to reduce the high prevalence, the most cost-effective of which were those that focused on the school environment. Although there is vast research that focus on interventions that address obesity through interventions to improve schoolchildren diets and physical activity level in many countries of the Latin American region, there is lack of evidence of the effectiveness of multicomponent interventions that aim to reduce the prevalence of obesity among schoolchildren in the Paraguayan context.

DETAILED DESCRIPTION:
Nutritional education and physical activity. Interventions that promote healthy eating and lifelong physical activity in schoolchildren through school programs aim to equip children with knowledge, attitudes and behavioral skills to help them establish and maintain a healthy lifestyle.

Poor diet quality has been identified as one of the main factors contributing to the obesity epidemic. Research has shown that a diet that includes the recommended servings of fruits and vegetables (VF) reduces morbidity and mortality from non-communicable diseases (NCDs) and has also been linked to a lower risk of adiposity. Therefore, the need to promote the consumption of VF from an early age through effective programs.

The interventions in Physical Activity have shown effective results in the decrease of BMI, the thickness of the skin folds and the percentage of fat mass in school-age children. Taking into account that currently the schoolchildren have decreased the amount of time dedicated to games, sports or other types of movement and the hours of sedentary life and in front of the screens (computers, tablets, television, mobile phones, others) have increased.

It is necessary to promote the performance of physical activity in the school environment through permanent programs that contribute to improving the physical condition of children, complying with daily recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Being public or private schools of the 22 districts of Caaguazú Department
* Having a minimum of 100 students in each of the three grades of second level of basic school education during 2017 school year
* Having physical education teachers

Exclusion Criteria:

* Schools that had only one school shift
* Schools that expressed their refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1568 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Skinfold thickness | 6 months
  Continuous variable, measured in millimeters (mm)

SECONDARY OUTCOMES:
Fruit and vegetables intake | 6 months
  Continuous variable, measured in servings per day
Physical activity level | 6 months
  Categorical variable, measured using MET in minutes/week and classified as low, medium and high intensity
Nutritional status | 6 months
  Categorical variable, measured using BMI/age an classified as undernourished, normal, overweight and obese according to WHO standards
Waist circumference | 6 months
  Continuous variable, measured in centimeters (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Rios, Study Director — IRIS UNCA
Locations (1):
- Instituto Regional de Investigacion en Salud, Coronel Oviedo, Caaguazú Department, Paraguay

IPD SHARING:
Plan to Share IPD: Yes
Protocol
Supporting Information: Study Protocol, SAP, ICF
Time Frame: all the time
Access Criteria: investigators